CLINICAL TRIAL: NCT01343589
Title: Effects of Milk Derived From Mountain-pasture Grazing Cows on Risk Markers of the Metabolic Syndrome Compared to Conventional Danish Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Dairy Research Foundation, Denmark (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Tine Tholstrup, Dpt Human Nutrition, University of Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-B-2009-052 (B del)
Record Dates: First submitted 2011-04-18; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Heart Disease; Type-2 Diabetes
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: milk fat — 39 g milk fat per day in 12 weeks
  Other Names: Yellow feed

SUMMARY:
To investigate the effect of milk delivered from mountain-pasture grazing cows on risk markers of the metabolic syndrome and type-2 diabetes with the effect of conventional Danish milk. The study should reveal the importance of phytanic acid content for these effects.

ELIGIBILITY:
Inclusion Criteria:

* sign written consent
* Age: 50-70
* BMI: 20-30
* increased risk of developing MS
* refrain from dietary supplements and blood donations prior to, and during the study

Exclusion Criteria:

* poor compliance
* if they suffering from any chronic or long lasting illness
* abuse of alcohol or medicine

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test | before and after the intervention (12 weeks)
LDL cholesterol | before and after the intervention (12 weeks)
HDL cholesterol | before and after the intervention (12 weeks)
Total cholesterol | before and after the intervention (12 weeks)
Triacylglycerol | before and after the intervention (12 weeks)
C-reactive protein | before and after the intervention (12 weeks)
fatty acid composition in plasma | before and after the intervention (12 weeks)

SECONDARY OUTCOMES:
phytanic acid | before and after the intervention (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, lector, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Werner LB, Hellgren LI, Raff M, Jensen SK, Petersen RA, Drachmann T, Tholstrup T. Effects of butter from mountain-pasture grazing cows on risk markers of the metabolic syndrome compared with conventional Danish butter: a randomized controlled study. Lipids Health Dis. 2013 Jul 10;12:99. doi: 10.1186/1476-511X-12-99. PMID 23842081